CLINICAL TRIAL: NCT03495232
Title: A Multicenter Prospective Cohort Study on Persona Total Knee System
Brief Title: Persona Cohort Nordic Multicenter Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: K.CR.I.EU.15.13 Cohort
Record Dates: First submitted 2018-03-20; First posted 2018-04-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Knee Arthropathy
Keywords: Total Knee Arthroplasty; Persona knee system; osteoarthrosis; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Zimmer Biomet Persona total knee system — Product manufactured by Zimmer Biomet used to replace the knee joint.

SUMMARY:
In this project the investigators wish to:

Evaluate intra-operative and postop complications, longer term survivorship and patient reported outcome measures (PROMs) following primary total knee replacement using Persona Total Knee system.

This project is carried out as prospective cohort study. Recruitment of participants to this project is expected to begin in October 2016 or as soon as permission from the Regional Ethics Committee and the local Data Protection Agency is obtained as required. A total of 700 participants (including 155 participants from a randomized controlled trial (RCT) investigating the Persona and the Nexgen total knee systems, which is separately submitted to the ethics committee) are to be included at several centers in the nordic region. Recruitment is expected complete after a period of 1,5 years per site. The patient follow-up visits are expected to be completed 2 years after recruitment of the last participant. Survivorship will be collected until 10 years after the recruitment of the last participant.

Participants are seen on an outpatient basis at 3 months and 1 and 2 years postoperatively.

After the 2 year follow-up visit the patients recruited in the Scandinavian sites will be followed for survivorship through the National Knee Arthroplasty Registries at 5, 7 and 10 years postoperatively. Since France does not have a national registry, the French site will also perform 5 year follow-up visits.

DETAILED DESCRIPTION:
The investigators will retain the subject data sources, case report forms (CRFs) and electronic-CRFs in accordance with local laws and regulations.

The enrollment is competitive between the participating centers. Project information and consent according to local requirements before surgery is completed.

Surgery is performed as described in the manufacturer's surgical technique. A senior surgeon dedicated to total knee arthroplasty surgery will perform all operations with an assistant.

Participants will receive standard pain treatment and rehabilitation until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological osteoarthritis of the knee set to receive a primary unilateral total knee replacement

Exclusion Criteria:

* Patients who are unwilling or unable to give consent, or to comply with the follow-up program.
* Patients that meet any contraindications listed in the Instruction for Use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient planned for primary total knee arthroplasty (TKA) on orthopedic surgeons' waiting list may be asked and selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2029-04-07 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate patient reported outcome measures following primary total knee replacement using Persona Total Knee system | 2 years
  Evaluate patient reported outcome measures following primary total knee replacement using Persona Total Knee system as measured by Oxford knee score (OKS); a 12-item patient-reported Patient Reported Outcomes specifically designed and developed to assess function and pain after total knee replacement surgery. Score ranging from 0 (most severe symptoms/problems) to 48 (least severe).

SECONDARY OUTCOMES:
Evaluate patient reported physical activity level following primary total knee replacement using Persona Total Knee system. An 8-item patient-reported outcome. Score ranging from 0 (most severe symptoms/problems) to 32 (least severe). | 2 years
  Oxford knee score Activity & Participation Questionnaire (OKS, APQ)
Evaluate patient quality of life following primary total knee replacement using Persona Total Knee system | 2 years
  EuroQol Group (EQ5D) standardized measure of health status. Measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Overall health status rated by the patient using the visual analogue scale (EQ-VAS).
Evaluate patient satisfaction following primary total knee replacement using Persona Total Knee system | 2 years
  Anchoring questions. Focusing on Patient perception of their knee and their satisfaction with the knee after their knee surgery
Evaluate patient reported awareness of their knee following primary total knee replacement using Persona Total Knee system | 2 years
  Forgotten Joint Score (FJS)
Evaluate intraoperative and postoperative complications | 10 years
  Register adverse events including intraoperative complications and revisions at any postoperative time point.
Evaluate implant positioning following primary total knee replacement using Persona Total Knee system | 2 years
  Measure radiolucency and osteolysis using conventional radiographs in anterior posterior (AP) and lateral views.
Evaluate longer term survivorship following primary total knee replacement using Persona Total Knee system | 10 years
  Survival of the implant through registries

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, Prof, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (4):
- Copenhagen University Hospital, Hvidovre, Copenhagen, Denmark
- Institute Locomoteur de L'Ouest, Saint-Grégoire, France
- St Olavs Hospital, Trondheim, Norway
- Ortopedic Clinic, Motala Specialist Care Capio AB, Motala, Sweden

IPD SHARING:
Plan to Share IPD: No